CLINICAL TRIAL: NCT06261840
Title: Refining Treatment Options for Trichomonas Vaginalis Infection in Women and Men: A Comparative Analysis of Oral Multi-Dose Metronidazole and Single-Dose Secnidazole
Brief Title: Refining Treatment Options for Trichomonas Vaginalis Infection: A Comparative Analysis of Metronidazole and Secnidazole
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: University of Alabama at Birmingham (Other); Louisiana State University Health Sciences Center in New Orleans (Other); Segal Trials Healthcare Clinical Data, Inc (Unknown)
Responsible Party: Principal Investigator, Patricia Kissinger, Principal Investigator, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-101
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Trichomonas Vaginitis; Bacterial Vaginitis
MeSH Terms: conditions — Trichomonas Vaginitis; Vaginosis, Bacterial | interventions — Metronidazole; secnidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Multi-Dose Metronidazole (Experimental): Multi-dose oral MTZ (500 mg twice daily for 7 days) for the treatment of T. vaginalis infection in women and men
  Interventions: Drug: Metronidazole 500 mg
- Single-Dose Secnidazole (Experimental): Single-dose 2 g oral SEC for the treatment of T. vaginalis infection in women and men
  Interventions: Drug: Secnidazole 2000 MG

INTERVENTIONS:
Drug: Metronidazole 500 mg — Multi-dose oral MTZ (500 mg twice daily for 7 days) for the treatment of T. vaginalis infection in women and men
  Other Names: FLAGYL
  Arms: Oral Multi-Dose Metronidazole
Drug: Secnidazole 2000 MG — Single-dose 2 g oral SEC for the treatment of T. vaginalis infection in women and men
  Other Names: SOLOSEC
  Arms: Single-Dose Secnidazole

SUMMARY:
This is a multi-centered, randomized, open-label, parallel, phase IV clinical trial comparing the effectiveness and cost-effectiveness of oral multi-dose metronidazole (MTZ) and oral single-dose secnidazole (SEC) for the treatment of Trichomonas vaginalis in both women and men.

DETAILED DESCRIPTION:
This is a multi-centered, randomized, open-label, parallel, phase IV clinical trial comparing the effectiveness and cost-effectiveness of oral multi-dose metronidazole (MTZ) and oral single-dose secnidazole (SEC) for the treatment of Trichomonas vaginalis in both women and men. The goal is to refine T. vaginalis treatment for women and men by examining the effectiveness (Aim 1) and cost-effectiveness (Aim 2) of multi-dose oral MTZ versus single-dose oral SEC. The investigators have several secondary analyses for Aim 1 including to examine if bacterial vaginosis (BV) interferes with T. vaginalis treatment, to explore preferences for follow-up visits, and to examine the natural history of T. vaginalis infection in both sexes.

If single-dose oral SEC is found to be superior to multi-dose oral MTZ, this could potentially result in an estimated 280,000 people in the U.S./year receiving better care, having fewer adverse sexual and reproductive health outcomes, and having a reduced risk for HIV acquisition. It will also provide patients with a single-dose oral treatment option that will be particularly attractive for subjects with concomitant T. vaginalis and BV.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18 years or older of any race/ethnicity will be included in the study.
* Participants must have either a positive T. vaginalis rapid antigen test (OSOM), or wet mount microscopy with motile trichomonads, or nucleic acid amplification test (NAAT) urinalysis or Pap smear positive for TV within two weeks of available results (and have not yet been treated) that is confirmed by repeat T. vaginalis NAAT testing at study enrollment,
* Willing and able to provide and understand informed consent to comply with the study protocol,
* Have a method of contact (either phone, email or social media),
* Be willing to be randomized.

Exclusion Criteria:

* Pregnant/lactating or seeking to be pregnant
* Have been treated for with a 5-nitroimidazole (i.e. Metronidazole (MTZ), tinidazole (TDZ), or secnidazole [SEC]) in the last 28 days
* Used intravaginal boric acid or any other intravaginal treatment for T. vaginalis in the last 14 days
* Have a history of a type 1 hypersensitivity reaction to 5-nitroimidazole medications
* Are taking phenytoin (Dilantin) and/or warfarin (Coumadin) due to drug-drug interactions with oral MTZ
* Use of medications which may alter the metabolism of MTZ including Lithium and barbiturates (amobarbital, butalbital, methohexital, phenobarbital, pentobarbital, primidone, secobarbital)
* Have been previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment, as Measured by the Number of Participants that are Cured of Trichomonas Vaginalis | A TOC visit will be scheduled 4 weeks (+- 1 week) after post completion of treatment
  A repeat T. vaginalis NAAT test will be completed at the test of cure (TOC) visit

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kissinger, PhD, Principal Investigator — Tulane University
Locations (4):
- United States (4):
  - University of Alabama at Birmingham [UAB] Gynecology Clinics, Birmingham, Alabama
  - UAB Sexual Health Research Clinic [SHRC], Birmingham, Alabama
  - Segal Trials Healthcare Clinical Data, Inc. 1065 NE 125th St. Suite 417 North Miami, FL 33161, North Miami, Florida
  - LSU-CrescentCare Sexual Health Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No